CLINICAL TRIAL: NCT06192719
Title: Establishment and Exploitation of a European-Latin American Research Consortium Towards Eradication of Preventable Gallbladder Cancer - EULAT Eradicate GBC
Brief Title: EULAT Eradicate GBC
Acronym: EULAT
Status: Recruiting | Type: Observational
Sponsor: Centre Paul Strauss (Other)
Collaborators: Heidelberg University Hospital (UKHD, Germany, Coordinator) (Unknown); Universidad Austral de Chile (UACH, Chile) (Unknown); Universidad de la Frontera (UFRO, Chile) (Unknown); Universidad Católica del Maule (UCM, Chile) (Unknown); Centre international de recherche sur le cancer (IARC, France) (Unknown); Universidad de Chile (UChile, Chile) (Unknown); Instituto Nacional de Enfermedades Neoplásicas (INEN, Peru) (Unknown); Universidad Mayor de San Simón (UMSS, Bolivia) (Unknown); Oslo University Hospital (Other); Sanatorio el Carmen (Argentina) (Unknown); Pontificia Universidad Católica de Chile (PUC, Chile) (Unknown); University of Bristol (Other); University of Oslo (Other); Chilean institutions (See detailed study description below) (Unknown); Peruvian institutions (See detailed study description below) (Unknown); Bolivian institutions (See detailed study description below) (Unknown); Argentinian institutions (See detailed study description below) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2023-020
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Gallbladder Cancer; Gallstone Disease
MeSH Terms: conditions — Gallbladder Neoplasms; Cholelithiasis | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Saliva, Urina, Bile, Feaces and Gallbladder tissue. Hemoderivatives (whole blood, serum, plasma and buffy coat).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gallbladder Cancer/Dysplasia: Patients affected by gallbladder cancer or dysplasia, both before and after starting their treatment
  Interventions: Other: None, observational study.
- Gallstone disease: Patients affected by cholelithiasis before cholecystectomy (only patients scheduled for cholecystectomy will be recruited)
  Interventions: Other: None, observational study.

INTERVENTIONS:
Other: None, observational study. — Epidemiological, clinical and dietary data will be collected along with blood, saliva, urine, bile, feces and gallbladder tissue samples.

SUMMARY:
Gallstones are relatively frequent in women and constitute one of the main risk factors for gallbladder cancer (GBC).

Currently, GBC diagnosis is mainly based on imaging (ultrasound or abdominal CT) associated with invasive examinations (biopsy and surgery), with no marker available to date to accurately predict risk and diagnose the disease early. The only curative treatment for GBC remains surgery with complete resection of tumors in early stages.

Given the aggressiveness of GBC and the very limited therapeutic options, as well as the possibility of preventing GBC by cholecystectomy during the 10 to 20 years required for the development of gallbladder tumors, it is imperative to develop effective and efficient prevention strategies based on a prioritization of interventions according to environmental and genetic-molecular risk factors.

The investigators aim to identify epidemiological factors linked to the development of GBC, and to identify, validate and functionally characterize genetic-molecular markers in blood, saliva, urine, bile and stool that allow risk prediction, early diagnosis and precision treatment of incidental tumors.

DETAILED DESCRIPTION:
Gallbladder cancer (GBC) is a neglected disease with huge potential for prevention. This study aims at significantly improving the accuracy of risk estimation and early detection of GBC by identifying and adequately considering geographical, environmental, lifestyle, ethnic, gender and molecular differences. The investigators plan to generate the information needed to establish and refine current prevention programmes, including the primary, secondary and tertiary prevention of GBC. The investigators will (1) build a unique European-Latin American GBC biorepository integrated into a tailored IT platform, (2) identify, validate and functionally characterize novel GBC biomarkers, (3) develop a multifactorial risk score that integrates established and newly identified epidemiological and molecular risk factors, (4) improve the understanding of the causal mechanisms that link lifestyle, cultural and behavioural factors to GBC development, (5) unravel novel opportunities for the targeted therapy of incidental GBC, (6) exploit existing and newly generated epidemiological and multi-omics data to improve the accuracy of GBC risk prediction and (7) contribute to the training of the next generation of Latin American researchers in precision medicine for GBC. The generated information will permit identification of individuals at high GBC risk, guiding surveillance and individual decisions on the possible benefit of preventive gallbladder removal in regions of low and high GBC incidence. Novel data on genomic alterations in incidental GBC will pave the way towards implementation of future clinical trials. The planned European-Latin American GBC biorepository and IT platform will constitute a prime resource for translational research on individualized prevention, personalized early detection and targeted therapy of GBC. The participation in our project of representatives of health authorities, patients and the industry guarantee the efficient incorporation of project results into national health policies.

The study protocol has been approved by the Comité de Protection des Personnes, France, the ethics committees of Servicio de Salud Metropolitano Oriente, Servicio de Salud Metropolitano Sur Oriente and Servicio de Salud Metropolitano Central in Santiago de Chile, Servicio de Salud Coquimbo in Coquimbo, Chile, Servicio de Salud Maule in Talca, Chile, Universidad Católica del Maule in Talca, Chile, Servicio de Salud Concepción in Concepción, Chile, Servicio de Salud Araucanía Sur in Temuco, Chile, Servicio de Salud Valdivia in Chile, Centro de Bioética Universidad del Desarrollo and Clínica Alemana de Santiago in Santiago de Chile, Unidad de Investigación Hospital San Juan de Dios in Santiago de Chile, the Medical Faculties of Universidad de Chile and Pontificia Universidad Católica de Chile, Facultad de Medicina, Universidad Mayor de San Simón, Bolivia, Comité Provincial de Ética de Investigación de la Provincia de Jujuy, Argentina, and Comité de ética e Investigación del Instituto Nacional de Enfermedades Neoplásicas, Peru.

ELIGIBILITY:
Inclusion Criteria:

1. Cohort A. Patients with gallbladder cancer or dysplasia, both before and after the start of their anticancer treatment.

   Cohort B. Patients with cholelithiasis before cholecystectomy (only patients scheduled for cholecystectomy will be recruited)
2. Diagnosis confirmed in accordance with standard protocols of the participating hospitals
3. Men and women aged 18 or over

Exclusion Criteria:

1. Any medical condition that present an unreasonable risk to the participant.
2. Any psychiatric condition that interferes with understanding informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are adults with GBC, gallbladder dysplasia, or cholelithiasis.
Sampling Method: Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Gallbladder Cancer/Dysplasia development | At inclusion or after pathological examination of the resected gallbladder

CONTACTS AND LOCATIONS:
Overall Officials: Justo LORENZO BERMEJO, PhD, Principal Investigator — Heidelberg University Hospital (UKHD, Germany) and Institut de cancérologie Strasbourg Europe (ICANS, France)
Locations (36):
- Argentina (3):
  - Hospital Papa Francisco, Salta
  - Sanatorio el Carmen, Salta
  - Hospital Pablo Soria, San Salvador de Jujuy
- Bolivia (5):
  - Complejo Hospitalario Viedma, Cochabamba
  - Hospital del Norte, Cochabamba
  - Hospital Obrero No. 2 (Caja Nacional del Seguro Social), Cochabamba
  - Instituto Gastroenterológico, Cochabamba
  - Instituto Oncológico Nacional, Cochabamba
- Chile (19):
  - Hospital Regional de Arica, Arica
  - Hospital Regional de Concepción, Concepción
  - Hospital De Puerto Montt, Port Montt
  - Hospital Clínico de Magallanes, Punta Arenas
  - Hospital Regional de Rancagua, Rancagua
  - Clínica Alemana de Santiago, Santiago
  - Fundación Arturo López Perez (FALP), Santiago
  - Hospital Barros Luco, Santiago
  - Hospital Clínico Universidad de Chile, Santiago
  - Hospital del Salvador, Santiago
  - Hospital El Pino, Santiago
  - Hospital Padre Hurtado, Santiago
  - Hospital San Borja, Santiago
  - Hospital San Juan de Dios, Santiago
  - Hospital Sótero del Río, Santiago
  - Hospital Regional de Talca, Talca
  - Clínica Alemana de Temuco, Temuco
  - Complejo Asistencial Padre Las Casas, Temuco
  - Hospital Regional de Temuco, Temuco
- Institut de cancérologie Strasbourg Europe, Strasbourg, France
- Peru (8):
  - Hospital Goyoneche, Arequipa
  - Hospital Honorio Delgado, Arequipa
  - Instituto Regional de Enfermedades Neoplásicas del Sur (IREN Sur), Arequipa
  - Clínica Monte Sinaí, Juliaca
  - Hospital Base III- La Capilla ESSALUD, Juliaca
  - Instituto Nacional de Enfermedades Neoplásicas (INEN), Lima
  - Hospital Regional Manuel Nuñez Butrón, Puno
  - Instituto Regional de Enfermedades Neoplásicas del Norte (IREN Norte), Trujillo

REFERENCES:
- See also: Related Info — http://www.SaludVesiculaBiliar.org